CLINICAL TRIAL: NCT02419963
Title: A New Dimension in Modeling Irritable Bowel Syndrome (IBS) to Elucidate Novel Diagnostic Biomarkers and Microbiome Signatures
Brief Title: Analyzing IBS to Identify Biomarkers and Microbiome Signatures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amy Foxx-Orenstein, PI, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14-008799
Record Dates: First submitted 2015-01-30; First posted 2015-04-17 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Diarrhoea Predominant Irritable Bowel Syndrome; IBS
Keywords: microbiome; biomarkers; Vitamin D; Serotonin
MeSH Terms: interventions — Endoscopy; Sigmoidoscopy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IBS-D patients (Other): Subjects on this arm will have an endoscopy for tissue biopsy, and provide blood samples and stool samples.
  Interventions: Procedure: endoscopy for tissue biopsy; Other: Blood Sample; Other: Stool Sample
- Healthy Controls (Other): Subjects on this arm will have an endoscopy for tissue biopsy, and provide blood samples and stool samples.
  Interventions: Procedure: endoscopy for tissue biopsy; Other: Blood Sample; Other: Stool Sample

INTERVENTIONS:
Procedure: endoscopy for tissue biopsy — endoscopy to obtain tissue biopsy for analysis of biomarker status
  Other Names: Sigmoidoscopy
Other: Blood Sample — Blood draw to evaluate serotonin and Vit D level.
Other: Stool Sample — Stool sample to evaluate microbiome fingerprint.

SUMMARY:
Microbiota from fecal samples from IBS-D patients, in combination with vitamin D supplementation added to our 3-D immunocompetent intestinal models will establish a high fidelity disease model to achieve our long-term goal to understand the relationship between gut microbiome, vitamin D levels, host gene expression and IBS-D symptoms that could ultimately be used as a testing platform for treatment and prevention.

DETAILED DESCRIPTION:
The pathophysiology of IBS is not well understood. Preliminary studies support IBS-D patients with varied microbiome fingerprints, vitamin D levels, and blood serotonin levels compared to non-IBS patients. The investigators have novel 3-D immunocompetent intestinal models to establish a new model of high fidelity disease to examine the relationship of IBS-D patients gut microbiome, with supplemental vitamin D levels, and the relationship of blood serotonin and vitamin D levels. IBS-D patients and healthy controls will be asked to provide a fecal sample, a biopsy sample of colonic tissue obtained during a clinically appropriate flexible sigmoidoscopy or colonoscopy, and a blood sample. There will be 1-2 office visits. One visit will last 30 minutes, the second visit no longer than 3 hours. This study is funded by a combined MAYO-Arizona State University seed grant. The samples will be analyzed at ASU. Our long-term goal is to understand the relationship between gut microbiome, vitamin D levels, host gene expression, serotonin levels, and IBS-D symptoms that could ultimately be used as a testing platform for treatment and prevention of this highly prevalent disorder.

ELIGIBILITY:
Inclusion criteria:

IBS-D subjects:

* Patients who fulfill IBS-D criteria, without causes of active inflammation.
* active symptoms for at least 2 months
* diagnosed at least 6 months prior to enrollment

Healthy Control:

- Healthy control patients should have no active infection or inflammation.

Exclusion criteria:

* does not meet inclusion criteria
* will not participate in blood draw, stool sample donation, or endoscopy
* history of acute illness within 3 months of testing
* any fecal transplant history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-12 (Actual)

PRIMARY OUTCOMES:
Serotonin level | Study Day 2
  2 blood vials will be drawn during the flexible sigmoidoscopy or colonoscopy procedure, and serotonin levels will be drawn from one of these blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Foxx-Orenstein, DO, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States